CLINICAL TRIAL: NCT05827640
Title: Determining Expiratory Time Constant in Mechanically Ventilated Patients
Brief Title: Expiratory Time Constant in Mechanically Ventilated Patients
Status: Completed | Type: Observational
Sponsor: East Slovak Institute for Cardiovascular Diseases (Other)
Responsible Party: Principal Investigator, Filip Depta MD, MD, East Slovak Institute for Cardiovascular Diseases
Other Study IDs: www.vusch.sk
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Comparing Six Different Methods to Obtain Expiratory Time Constant
Keywords: expiratory time constant, mechanical ventilation, exhalation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data recording using conventional ventilation strategies (PCV and VCV) — no intervention

SUMMARY:
Determining expiratory time constants in mechanically ventilated patients

DETAILED DESCRIPTION:
Adult patients (n = 30) undergoing elective cardiac surgery with extracorporeal circulation (ECC) were included. Patients were excluded from the study if they had any known lung disease or had previous thoracic surgery. After the surgery, all patients were transferred to the intensive care unit (ICU) and connected to well-established Servo-U (Maquet, Getinge AB, Solna, Sweden) mechanical ventilator. First, the ventilation mode was set to mandatory volume-controlled ventilation (VCV) for 15 minutes. After that, mandatory pressure-controlled ventilation (PCV) for another 15 minutes was commenced. All patients were in supine position, sedated and paralyzed using continuous infusion of propofol and atracurium with no spontaneous breathing efforts. During VCV, an end-inspiratory pause (TPAUSE 10%) has been added to obtain inspiratory plateau pressure (P PLAT) under static conditions. Respiratory variables in VCV for all patients were as follows: PEEP 6 - 9 cmH 2 O depending on the local protocol, protective tidal volume (Vt) of 7 ml/kg/PBW, T PAUSE was set to 10%, I:E ratio of 1:2, rise time 5% and the respiratory rate was 14 breaths/min. After 15 minutes, VCV was changed to PCV with the same ventilator setting with inspiratory pressure set in the way to best match the Vt during the VCV. ARDSNet tables were used to determine PBW for all patients.

A novel device enabling data acquisition (Dr. Wave, Quadrus Medical Technologies, NY, White Plains, USA) has been connected to the Servo-U ventilator after admission to the ICU to record flow, pressure, and volume waveforms. All data in the study were derived from measurements and calculations from this device and included: Peak Inspiratory Pressure (PIP), PPLAT, PEEP, expiratory tidal volume (Vt) respiratory system compliance (C RS ), airway resistance (RTOT) and the peak expiratory flow rate (PEFR).

Based on obtained data of flow, volume and pressure during PCV and VCV, six different methods to determined expiratory time constant were examined

ELIGIBILITY:
Inclusion Criteria: cardiac surgery with extracorporeal circulation

-

Exclusion Criteria:

* known pulmonary disease
* previous thoracic surgery
* poor preoperative cardiac status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiac surgery with extracorporeal circulation (mostly CABG or AVR).
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Expiratory time constant | 3 months
  Six different methods to assess expiratory time constants in mechanically ventilated patients

SECONDARY OUTCOMES:
Validity of expiratory time constant definition | 3 months
  To prove if three time constant correspond to actual first time constant multiplied by the factor of 3

CONTACTS AND LOCATIONS:
Overall Officials: Dušan Rybár, PhD, Study Director — East Slovak Institute for Cardiovascular Diseases
Locations (1):
- East Slovak Institute for Cardiovascular Diseases, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided